CLINICAL TRIAL: NCT06260735
Title: Non-invasive Spinal Cord Stimulation for Improving Movement: Neuromodulation With Spinal Stimulation Methods and Individualized Locomotor Training
Brief Title: Non-invasive Spinal Cord Stimulation After Spinal Cord Injury
Acronym: SCI-ES-WALK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Katinka Stecina, Associate Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS25897 (H2023:073); URGP#51472 (Other Grant/Funding Number: University of Manitoba); RGPIN-2015-05703 (Other Grant/Funding Number: NSERC)
Record Dates: First submitted 2023-11-28; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases
Keywords: Trans-spinal electrical stimulation; Locomotor training; Functional electrical stimulation; Peripheral nerve stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treadmill training combined with muscle and spinal cord stimulation (Experimental): Locomotor training is defined as walking on a treadmill with appropriate bodyweight support and augmented with muscle activation either by electrical nerve or muscle stimulation based on individual needs. Then, spinal stimulation will be integrated during training with on/off bouts alternating.
  Interventions: Device: Trans-spinal electrical stimulation; Device: Electrical muscle activation; Other: Treadmill walking

INTERVENTIONS:
Device: Trans-spinal electrical stimulation — Trans-spinal electrical stimulation (ts-ES) at T11-L1 vertebral levels with short pulses at a set frequency (30Hz).
Device: Electrical muscle activation — Peripheral nerve (PN) or muscle (NMES) stimulation strategy was developed for each participant to optimize stance/walk capacity based on personal needs/preferences.
Other: Treadmill walking — Stepping on a treadmill with individually preferred speed.

SUMMARY:
Spinal cord injury (SCI) is a central nervous system injury that often leads to motor dysfunction. Non-invasive electrical stimulation of the spinal cord has been recognized as a potential method of reactivating lost spinal neural networks to improve motor recovery and exercise response after SCI. Trans-spinal electrical stimulation (ts-ES) has been found to increase functional gains in people after SCI when applied in combination with other motor training protocols.

This project aims to evaluate the effects of non-invasive lumbar spinal cord electrical stimulation on the motor function of trunk and lower limbs in people with SCI after augmenting their locomotor training (treadmill stepping) with step-cycle-based electrical peripheral neural stimulation methods.

DETAILED DESCRIPTION:
This project will evaluate the effects of non-invasive lumbar ts-ES on locomotor function in people with incomplete motor SCI (iSCI) who retain some ability to stand or walk.

This study has 3 phases:

Baseline assessment - 2 sessions - week 1 -Lab visits #1-2

Locomotor training with varied electrical stimulation- 12 sessions - weeks 2-5 - Lab visits #3-14 (1hr, x3/week)

End of training assessment - 2 sessions - week 6- Lab visits #15-16.

Specific locomotor deficits of each participant will be evaluated, and their step-cycle-based peripheral muscle or nerve stimulation strategy will be determined accordingly to improve stance or step capacity. After augmenting their locomotor function with muscle or peripheral nerve stimulation-induced activation strategies that address particular and unique motor deficits, they will receive intermittent bouts of stance or locomotor training supplemented with ts-ES. The locomotor training will consist of standing/walking on a treadmill with appropriate bodyweight support and added muscle or peripheral nerve stimulation.

Specifically, the project aims to assess the following:

1. Does combined muscle (NMES) or peripheral nerve (PN) stimulation with ts-ES during treadmill stepping facilitate locomotor performance?
2. Does four weeks of combined training as described above (1hrx3/week) facilitate exercise capacity (measured by submaximal VO2) in persons with chronic iSCI?

ELIGIBILITY:
Inclusion Criteria:

* Has spinal cord injury, 6 mo or longer since injury
* Is between 20 and 65 years of age
* Has difficulty with trunk and/or lower limb function
* Stable medical condition
* Non-progressive etiology of spinal injury
* No ventilatory support

Exclusion Criteria:

* Genetic or degenerative etiology of spinal injury
* Need for ventilatory or other life-sustaining medical support
* History of cardiovascular or pulmonary complications (heart failure, severe hypertension etc.)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Neurophysiological markers or stepping | Pre-training (on week 1) and within one week from end of training (on week 6)
  Average step length, step height at ankle (cm).
Electromyography (EMG) of ankle extensor muscles | Pre-training (on week 1) and within one week from end of training (on week 6)
  Mean RMS amplitude
Metabolic function testing | Pre-training (on week 1) and within one week from end of training (on week 6)
  Breath-by-breath analysis of air in/out will be used to measure VO2max (mL/kg/min).

SECONDARY OUTCOMES:
6 Min Walk Test | Pre-training (on week 1) and within one week from end of training (on week 6)
  Measure distance (m) covered in 6 min walking, overground with device of choice (if using it at home/in community). Repeat with save device. Verbal encouragement and safety support in place during testing.
SCIM-Spinal Cord Independence Measure- Mobility scores | Pre-training (on week 1) and within one week from end of training (on week 6)
  Rick Hansen Institute, Spinal Cord Independence Measure III - Mobility subsection, Questions 12-17. Scale: 0-20. Lower score means less mobility.
Autonomic scores | Pre-training (on week 1) and within one week from end of training (on week 6)
  American Spinal Injury Association-Autonomic Standards assessment form-General Autonomic Function & Lower Urinary tract, bowel, and sexual function components. Scale: 0-48. Lower scores mean less autonomic function.
Rate or Perceived Exertion (RPE) of Submaximal VO2 testing | Pre-training (on week 1) and within one week from end of training (on week 6)
  Borg scale from 6-20 (chart used from Heart Online open source). Scale: 6-20. Lower scores mean less exertion (less tiring).

CONTACTS AND LOCATIONS:
Overall Officials: Katinka Stecina, Principal Investigator — University of Manitoba; Kristine Cowley, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No